CLINICAL TRIAL: NCT06662175
Title: Role of Dexmedetomidine as Synergistic Agent to Prolong a Subarachnoid Block Duration
Brief Title: Role of Dexmedetomidine as Synergistic Agent
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Responsible Party: Principal Investigator, Faryal Uzma, Faryal Uzma Prinicipal Investigator, Lady Reading Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 359/LRH/MTI
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Dexmedetomidine; Hyperbaric Bupivacaine; Subarachnoid Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A Hyperbaric Bupivicaine (Experimental): Group A (Unexposed) will received 2 ml of intrathecal bupivacaine.
  Interventions: Drug: Hyperbaric bupivacaine
- GROUP B Hyperbaric Bupivacaine and Dexmedetomidine (Experimental): Group B (Exposed) will receive a combination of bupivacaine and Dexmedetomidine infusion.
  Interventions: Drug: hyperbaric bupivacaine and dexmedetomidine

INTERVENTIONS:
Drug: Hyperbaric bupivacaine — Group A (Unexposed) will received 2 ml of intrathecal bupivacaine
  Arms: Group A Hyperbaric Bupivicaine
Drug: hyperbaric bupivacaine and dexmedetomidine — Group B (Exposed) will receive a combination of bupivacaine and Dexmedetomidine infusion
  Arms: GROUP B Hyperbaric Bupivacaine and Dexmedetomidine

SUMMARY:
The aim of this clinical trial is to contribute valuable insights into the role of Dexmedetomidine as a synergistic agent in prolonging subarachnoid block duration, with the overarching goal of enhancing perioperative care and surgical success rates.

DETAILED DESCRIPTION:
Dexmedetomidine is a frequently used alpha-2 adrenergic agonist for anesthesia and sedation due to its excellent selectivity. Dexmedetomidine can cause drowsiness, analgesia, and sympathetic reactions when injected intravenously. Dexmedetomidine has been investigated for possible synergistic benefits when used in conjunction with hyperbaric bupivacaine for subarachnoid block, sometimes referred to as spinal anesthesia. Because hyperbaric bupivacaine can produce a rapid onset and a longer duration of sensory and motor blockage, it is a common local anesthetic used in spinal anesthesia.

Numerous research studies have examined the synergistic effects of intravenous dexmedetomidine and hyperbaric bupivacaine in subarachnoid blocks. These effects are primarily observed in terms of extending the duration of sensory and motor blockade, enhancing postoperative analgesia, decreasing intraoperative and postoperative opioid consumption, and improving patient satisfaction. The mechanism underlying this synergistic effect is believed to be connected to the effects of dexmedetomidine on the central nervous system, which include its capacity to modify pain pathways, improve spinal anesthesia, and produce drowsiness and anxiolysis.

Although the combination of dexmedetomidine with hyperbaric bupivacaine has demonstrated encouraging outcomes in a number of studies, there is still discussion and continuing research over the best time, dosage, and patient selection criteria. As with any anesthesia procedure, the best course of action should be determined after taking into account specific patient considerations such age, comorbidities, and concurrent drugs.

Hameed et al compare the Synergistic effect of Dexmedetomidine on Subarachnoid Block with Hyperbaric Bupivacaine among three groups. In there study Patients in Group 1 received 2 ml of intrathecal bupivacaine; Group 2 received a combination of bupivacaine and Dexmedetomidine infusion; and Group 3 received bupivacaine followed by Dexmedetomidine infusion. Their study show that onset time of sensory blockade. The duration of sensory blockade and the rate of recovery of complete sensory block was significantly higher in Group 2 compared to Group 1. The distribution of adverse effect among group 1 and group 2 was, hypotension 20% vs 40%, Bradycadria 8% vs 24%, and Nausea 12% vs 12% respectively.

Previous studies have indicated that Dexmedetomidine can enhance the duration and quality of sensory blockade, improve postoperative analgesia, and reduce opioid consumption when used in conjunction with hyperbaric bupivacaine. Despite these promising findings, further exploration is warranted to elucidate the optimal dosage, timing, and patient selection criteria for Dexmedetomidine administration in subarachnoid blocks. Understanding the mechanistic basis of Dexmedetomidine's synergistic effects on subarachnoid block duration is crucial for refining anesthesia protocols and ultimately improving patient outcomes. By conducting this research study, the investigators aim to contribute valuable insights into the role of Dexmedetomidine as a synergistic agent in prolonging subarachnoid block duration, with the overarching goal of enhancing perioperative care and surgical success rates.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender aged between 18 and 65 years.
2. Patients scheduled for surgical procedures of lower limb requiring subarachnoid anesthesia.
3. American Society of Anesthesiologists (ASA) physical status classification I or II.

Exclusion Criteria:

1. Patients with contraindications to subarachnoid anesthesia, including severe coagulopathy, infection at the site of injection, or increased intracranial pressure.
2. Patients with a history of significant cardiac, respiratory, hepatic, or renal disease.
3. Pregnant or lactating women.
4. Patients with a history of substance abuse or dependence.
5. Patients on chronic opioid therapy or with opioid tolerance.
6. Patients with neurological deficits affecting sensation or motor function in the lower extremities.
7. Patients with psychiatric disorders affecting their ability to cooperate during the procedure or follow instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of Dexmedetomidine when used adjunctively with hyperbaric bupivacaine in extending the duration of sensory and motor blockade in subarachnoid anesthesia. | periodically motor blockade will be assessed until the achievement of modified Bromage score 3 from giving anesthesia till shifting of the patient to parent ward
  Sensory Blockade Duration: This refers to the time interval from the administration of the subarachnoid block until the complete recovery of sensory function in the dermatomes affected by the anesthesia. It will be assessed using standardized sensory tests, such as pinprick or cold sensation, within the affected dermatomes.
  Motor Blockade Duration:It encompasses the time from the onset of motor blockade to the complete recovery of motor function and will assessed by evaluating muscle strength and movement capability using modified Bromage score as
  0=Subject is able to lift the leg straight and move the hip, knee and ankle.
  1. Subject is unable to lift the leg straight but is able to lift the leg straight but is able to flex the knee and ankle freely.
  2. Subject is unable to flex the knee and hip, but is able to flex the ankle.
  3. Subject is unable to flex the ankle, knee, and hip, but is able to move toes.
  4. No movement in the lower extremity.

SECONDARY OUTCOMES:
Investigate the safety profile of Dexmedetomidine in combination with hyperbaric bupivacaine, in term of adverse events such as hypotension, bradycardia, and patient satisfaction. | till the shifting of patient to parent ward.
  Sedation levels will be assessed using the Ramsay score
  1. Awake; agitated or restless or both
  2. Awake; cooperative, oriented, and tranquil
  3. Awake but responds to commands only
  4. Asleep; brisk response to light glabellar tap or loud auditory stimulus
  5. Asleep; sluggish response to light glabellar tap or loud auditory stimulus
  6. Asleep; no response to glabellar tap or loud auditory stimulus Adverse Event: will be measured in following term Hypotension: defined as a systolic blood pressure less than 90 mm Hg or a mean arterial pressure below 60 mm Hg.
  Bradycardia:defined as a heart rate of less than 50 beats per minute. Patient Satisfaction:defined in terms of subjective assessment of the patient's physical and emotional well-being during the procedure include observed signs of distress, facial expressions, and verbal feedback. Patients' satisfaction will be assessed using a 10cm Visual Analogue Score. Where 10cm denoted maximal satisfaction and 0cm denoted minimal.

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Reading Hospital Mti Peshawar Kp Pakistan, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
the patients identity will be kept anonymous

REFERENCES:
- [Background] Sharma A, Varghese N, Venkateswaran R. Effect of intrathecal dexmedetomidine versus intravenous dexmedetomidine on subarachnoid anesthesia with hyperbaric bupivacaine. J Anaesthesiol Clin Pharmacol. 2020 Jul-Sep;36(3):381-385. doi: 10.4103/joacp.JOACP_323_17. Epub 2020 Sep 14. PMID 33487907